CLINICAL TRIAL: NCT02954172
Title: Study to Evaluate the Efficacy and Safety of IBI305 in Combination With Paclitaxel/Carboplatin Versus Bevacizumab in Combination With Paclitaxel/Carboplatin in Treatment-naïve Patients With Advanced or Recurrent Non-squamous NSCLC
Brief Title: Evaluate the Efficacy and Safety of IBI305 in Patients With Advanced or Recurrent Non-squamous NSCLC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Collaborators: WuXi CDS Clinical Research (Shanghai) Co.Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI305A301
Record Dates: First submitted 2016-10-23; First posted 2016-11-03 (Estimated); Results first posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-11

CONDITIONS: NSCLC
MeSH Terms: interventions — Bevacizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bevacizumab in Combination With Paclitaxel/Carboplatin (Experimental): Drug Bevacizumab15mg/kg in combination with Paclitaxel/Carboplatin 6 cycles then maintains at 7.5 mg/kg
  Interventions: Drug: Bevacizumab in Combination With Paclitaxel/Carboplatin
- IBI305 in Combination with Paclitaxel/Carboplatin (Active Comparator): Drug IBI305 15mg/kg in combination with Paclitaxel/Carboplatin 6 cycles then maintains at 7.5 mg/kg
  Interventions: Drug: IBI305 in Combination with Paclitaxel/Carboplatin

INTERVENTIONS:
Drug: Bevacizumab in Combination With Paclitaxel/Carboplatin — Drug Bevacizumab15mg/kg in combination with Paclitaxel/Carboplatin 6 cycles then maintains at 7.5 mg/kg
  Other Names: Avastin
  Arms: Bevacizumab in Combination With Paclitaxel/Carboplatin
Drug: IBI305 in Combination with Paclitaxel/Carboplatin — Drug IBI305 15mg/kg in combination with Paclitaxel/Carboplatin 6 cycles then maintains at 7.5 mg/kg
  Other Names: Bevacizumab Biosimilar
  Arms: IBI305 in Combination with Paclitaxel/Carboplatin

SUMMARY:
A randomized, double blind, multicenter phase3 study .

DETAILED DESCRIPTION:
A randomized, double blind, multicenter phase3 study in chemotherapy naive patients with stage IIIB,IV or recurrent NSCLC of non-squamous. the study will randomize about 436 patients at a 1:1 ratio to 2 treatment arms. The study is divided 4 phase, screening, combination treatment, maintenance and follow up.

ELIGIBILITY:
Inclusion Criteria:

1. signed inform consent form(ICF)
2. Age ≥ 18 years and ≤ 75 years, male or female
3. Histologically or cytologically documented inoperable, local advanced (stage IIIB), metastatic (stage IV), or recurrent non-squamous NSCLC; Mixed tumors should be categorized according to the predominant cell type
4. Histologically confirmed epidermal growth factor receptor (EGFR) wild type or insensitive mutation
5. At least one measurable lesion according to Response Evaluation Criteria In Solid Tumors（RECISIT） v 1.1
6. Eastern Cooperative Oncology Group(ECOG) performance status of 0 or 1
7. Life expectancy ≥ 6 months
8. Laboratory results:

   1. Adequate hematologic function, defined as absolute neutrophil count ≥1.5×10^9 /L, platelet count ≥100 ×10^9 /L, hemoglobin ≥90g/L;
   2. Adequate liver function, defined as total bilirubin levels ≤ 1.5 times normal upper limit (ULN), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 times ULN, or AST and ALT levels ≤ 5 times ULN for patients with hepatic metastasis;
   3. Adequate renal function, defined as serum creatinine ≤ 1.5 times ULN or creatinine clearance ≥ 50 ml / min (Cockcroft-Gault formula) and proteinuria < 2+;
   4. Coagulation function is adequate, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times normal upper limit (ULN), PTT or aPTT ≤ 1.5 times ULN;
9. Expected protocol compliance
10. Patients of childbearing potential must agree to use effective contraceptive measures during study treatment and for 6 months after receiving last study treatment (e.g. abstinence, sterilization surgery, oral contraceptives, contraception by progesterone injection or subcutaneous).

Exclusion Criteria:

1. Prior chemotherapy or target therapy with another systemic anti-cancer agent (e.g., monoclonal antibody, tyrosine kinase inhibitor) for the treatment of the patient's current stage of disease (Stage IIIB not amenable for combined modality treatment, stage IV or recurrent disease). Prior surgery and irradiation is permitted, provided that the criteria outlined in the protocol for both treatments are met. Disease progressed within 6 months after adjuvant therapy must be excluded.
2. Mixed non-small cell and small cell carcinoma, or mixed adenosquamous carcinomas with predominant squamous cell
3. Histologically or cytologically confirmed EGFR sensitive mutation type, unknown EGFR status for any reason is allowed in this study.
4. Known hemoptysis within 3 months prior to screening with blood volume more than 2.5 mL each time
5. Evidence of tumor invading major blood vessels on imaging. The investigator or the local radiologist must exclude evidence of tumor that is fully contiguous with, surrounding, or extending into the lumen of a major blood vessel (e.g., pulmonary artery or superior vena cava)
6. Evidence of brain metastasis, spinal cord compression or carcinomatous meningitis history with clinical symptoms. For stable patients with no symptom, could be admitted if fulfill all below criteria: measurable lesion(s) out of CNS, no metastasis at mesocephalon, annular protuberance, medulla oblongata and spinal cord; no history of intracranial bleeding.
7. Radical radiotherapy to the thorax with curative intent within 28 days prior to enrollment; palliative radiotherapy for bone lesions outside the thoracic region within 2 weeks prior to first dose of study treatment.
8. Serious, non-healing wound, active ulcer, or untreated bone fracture, or major surgical procedure within 28 days prior to randomization or anticipation of need for major surgery during the course of the study.
9. Minor surgery (Including insertion of an indwelling catheter) within 48 hours prior to first dose of study treatment
10. Recent or current (within 10 days prior to first dose of study treatment) receive treatment of Aspirin (> 325 mg/day) or other non-steroidal anti-inflammatory drugs (NSAID) known to inhibit platelet function (within 10 days prior to first dose of study treatment)
11. Recent or current receive treatment of oral all doses of oral or parenteral anticoagulants or thrombolytic agent. Prophylactic use of anticoagulants is permitted.
12. History or evidence of inherited bleeding diathesis or coagulopathy or thrombus
13. Uncontrolled hypertension (SBP>140 mmHg and/or diastolic blood pressure>90 mmHg), prior history of hypertensive crisis and hypertensive encephalopathy
14. Clinically significant cardiovascular disease but not limited to active infections; unstable angina; stroke or transient cerebral ischemia (within 6 months prior to screening); myocardial infarction (within 6 months prior to screening) ; congestive heart-failure (New York Heart Association (NYHA) class≥ II) ; serious cardiac arrhythmia, hepatic, renal or metabolic disease requiring medication during the study.
15. History of peptic ulcer, gastrointestinal perforation, erosive esophagitis, erosive gastritis, inflammatory bowel disease or diverticulitis, abdominal fistula or intra-abdominal abscess within 6 months prior to screening
16. Patient diagnosed with a tracheo-esophageal fistula
17. Clinically significant third space effusion (e.g., uncontrolled ascites or pleural effusion by extraction or other treatment)
18. Pulmonary fibrosis or active pneumonia showed by CT at baseline
19. Active malignancy other than non-small cell lung cancer (NSCLC), treated carcinoma in situ of the cervix, superficial basal cell or squamous cell carcinoma, radical surgery of localized prostate cancer, radical surgery of ductal carcinoma in situ within 5 years prior to randomization
20. Known autoimmune disease
21. Known positive HbsAg and hepatitis B virus (HBV)-DNA drop test in peripheral blood ≥ 1 x 10^3 copy number/L or 200 IU/mL; If HBsAg positive and HBV-DNA drop test in peripheral blood < 1 x 10^3 copy number/L or 200 IU/mL, patient is considered to be eligible by investigator only when chronic hepatitis B in the plateau and do not increase the risk
22. Known positive HIV or hepatitis C virus (HCV) or syphilis
23. Known allergic disease or allergic physique
24. Treatment with any other investigational agent or participation in another clinical trial within 30 days prior to screening
25. Known alcoholism or drug abuse
26. Pregnant or anticipation of pregnant during the study or lactating women
27. Known hypersensitivity to bevacizumab or any of its excipients and/or any of the chemotherapy agents
28. Other conditions that the investigator thinks unsuitable in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2019-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center; Sun Yat sen University;, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang Y, Wu B, Huang L, Shi M, Liu Y, Zhao Y, Wang L, Lu S, Chen G, Li B, Xie C, Fang J, Yang N, Zhang Y, Cui J, Song Y, Zhang C, Mei X, Cao B, Yang L, Cheng Y, Ying K, Sun T, Ren B, Yu Q, Liao Z, Pei Z, Wang M, Zhou J, Yu S, Feng G, Wan H, Wang H, Gao S, Wang J, An G, Geng Y, Ji Y, Yuan Y, Ma S, Jia Z, Hu M, Zhou H, Yu J, Sun X, Zhang L. Biosimilar candidate IBI305 plus paclitaxel/carboplatin for the treatment of non-squamous non-small cell lung cancer. Transl Lung Cancer Res. 2019 Dec;8(6):989-999. doi: 10.21037/tlcr.2019.12.23. PMID 32010577

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab in Combination With Paclitaxel/Carboplatin | IBI305 in Combination With Paclitaxel/Carboplatin
Started | 226 | 224
Completed | 220 | 221
Not Completed | 6 | 3
Not completed — Protocol Violation | 3 | 0
Not completed — allergic reaction | 2 | 1
Not completed — non-measurable lesions at baseline | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab in Combination With Paclitaxel/Carboplatin | IBI305 in Combination With Paclitaxel/Carboplatin | Total
Number analyzed (Participants) | 220 | 221 | 441
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean (SD) | 57.6 (8.69) | 57.2 (9.28) | 57.4 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 79 | 162
  Male | 137 | 142 | 279
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han | 217 | 211 | 428
  Others | 4 | 9 | 13
Region of Enrollment [Number; unit: participants]
  China | 220 | 221 | 441
Height [Mean (Standard Deviation); unit: centimeter] | 164.93 (8.166) | 164.03 (7.829) | 164.48 (8.003)
Weight [Mean (Standard Deviation); unit: kilogram] | 62.16 (10.844) | 62.14 (10.272) | 62.15 (10.550)

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: ORR（objective response rate）was defined as the percentage of participants in the analysis population who had a Complete Response or a Partial Response per RECIST 1.1. The percentage of participants who experienced a CR or PR is presented. Overall Response (OR) = CR + PR.
Time Frame: 18 weeks
Measure: Number; unit: percentage of participants
Groups:
- Bevacizumab in Combination With Paclitaxel/Carboplatin: Drug Bevacizumab 15mg/kg in combination with Paclitaxel/Carboplatin 6 cycles then maintains at 7.5 mg/kg
Arm/Group | Bevacizumab in Combination With Paclitaxel/Carboplatin | IBI305 in Combination With Paclitaxel/Carboplatin
Number analyzed (Participants) | 220 | 221
percentage of participants | 46.4 | 44.3
Statistical Analysis 1: Comparison: Bevacizumab in Combination With Paclitaxel/Carboplatin vs IBI305 in Combination With Paclitaxel/Carboplatin; Test type: Equivalence — the equivalence margin of the ORR ratio was set at (0.75, 1.33); Odds Ratio (OR) = 0.90, 90% CI 2-sided [0.756 to 1.077]

2. Secondary Outcome: Overall Survival Time
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: 18.020 months
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Bevacizumab in Combination With Paclitaxel/Carboplatin | IBI305 in Combination With Paclitaxel/Carboplatin
Number analyzed (Participants) | 220 | 221
month | NA [NA to NA] — insufficient number of participants with events | 18.020 [16.73 to NA] — insufficient number of participants with events
Statistical Analysis 1: Comparison: Bevacizumab in Combination With Paclitaxel/Carboplatin vs IBI305 in Combination With Paclitaxel/Carboplatin; Test type: Equivalence; p = 0.7066, Log Rank

3. Secondary Outcome: Progression-free Survival
Description: Progression-Free Survival (PFS) Per RECIST 1.1 as Assessed by Independent Radiological Review Committee.Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- IBI305 in Combination With Paclitaxel/Carboplatin: Drug IBI30515mg/kg in combination with Paclitaxel/Carboplatin 6 cycles then maintains at 7.5 mg/kg
Arm/Group | Bevacizumab in Combination With Paclitaxel/Carboplatin | IBI305 in Combination With Paclitaxel/Carboplatin
Number analyzed (Participants) | 220 | 221
months | 8.260 [6.810 to 8.500] | 8.430 [7.170 to 9.590]
Statistical Analysis 1: Comparison: Bevacizumab in Combination With Paclitaxel/Carboplatin vs IBI305 in Combination With Paclitaxel/Carboplatin; Test type: Equivalence; p = 0.3497, Log Rank

ADVERSE EVENTS:
Time Frame: through study completion, an average of 2 year
Arm/Group | Bevacizumab in Combination With Paclitaxel/Carboplatin | IBI305 in Combination With Paclitaxel/Carboplatin
All-Cause Mortality (participants affected / at risk) | 5/226 | 6/224
Serious Adverse Events (participants affected / at risk) | 85/226 | 75/224
Other Adverse Events (participants affected / at risk) | 222/226 | 216/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab in Combination With Paclitaxel/Carboplatin (N=226) | IBI305 in Combination With Paclitaxel/Carboplatin (N=224)
Lung infection (Infections and infestations) | 7 | 11
Pneumonia (Infections and infestations) | 3 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 4
Anaemia (Blood and lymphatic system disorders) | 8 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Vomiting (Gastrointestinal disorders) | 4 | 0
Fever (General disorders) | 3 | 2
Platelet count decreased (Investigations) | 27 | 24
White blood cell count decreased (Investigations) | 10 | 7
Neutrophil count decreased (Investigations) | 13 | 6
pulmonary infection (Infections and infestations) | 7 | 11
Infectious Pneumonia (Infections and infestations) | 3 | 3
upper respiratory infection (Infections and infestations) | 3 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
pharyngitis (Infections and infestations) | 0 | 1
urinary tract infection (Infections and infestations) | 0 | 1
gastroenteritis (Infections and infestations) | 1 | 1
Device associated infection (Infections and infestations) | 0 | 1
Fever infection (Investigations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
The anus infection (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Phthisis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0
Central nervous system metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
lymphangitis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 8 | 4
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 2
Anaphylaxis occurs almost instantaneously (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Hypoproteinemia (Metabolism and nutrition disorders) | 0 | 1
hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Reduced food intake (Metabolism and nutrition disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 2 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 1
Cerebrovascular disorders (Nervous system disorders) | 0 | 1
Cerebral hemorrhage (Nervous system disorders) | 1 | 0
Neurophlegmon (Nervous system disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Angle-closure glaucoma (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 0 | 1
Meibomianitis (Eye disorders) | 1 | 0
Retinal hemorrhage (Eye disorders) | 1 | 0
Congestive heart-failure (Cardiac disorders) | 0 | 2
Ventricular premature contraction (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 2
Myocardial infarction (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0
Wolfe-parkinson-white syndrome (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Hydropericardium (Cardiac disorders) | 1 | 0
Distal embolization (Vascular disorders) | 0 | 1
Limb vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Bronchorrhagia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Breathing difficulties (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Expectoration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Emesis (Gastrointestinal disorders) | 4 | 0
Esophageal obstruction (Gastrointestinal disorders) | 1 | 0
Saprodontia (Gastrointestinal disorders) | 1 | 0
Hepatic disease (Hepatobiliary disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Gout joint inflammation (Musculoskeletal and connective tissue disorders) | 1 | 0
Fever (Product Issues) | 3 | 2
death (Product Issues) | 0 | 2
Debilitation (Product Issues) | 0 | 1
Decreased platelet count (Investigations) | 27 | 24
Lower white blood cell count (Investigations) | 10 | 7
Neutrophils count decreased (Investigations) | 13 | 6
Alanine aminotransferase is elevated (Investigations) | 1 | 2
Aspartate aminotransferase was elevated (Investigations) | 1 | 2
Gamma-glutamyl transferase is elevated (Investigations) | 0 | 1
Haemoglobin reduction (Investigations) | 1 | 0
Blood bilirubin is elevated (Investigations) | 1 | 0
Tracheorrhagia (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab in Combination With Paclitaxel/Carboplatin (N=226) | IBI305 in Combination With Paclitaxel/Carboplatin (N=224)
Upper respiratory tract infection (Infections and infestations) | 21 | 23
Anaemia (Blood and lymphatic system disorders) | 54 | 53
decreased appetite (Metabolism and nutrition disorders) | 18 | 18
Hypokalemia (Metabolism and nutrition disorders) | 11 | 17
Sleeplessness (Psychiatric disorders) | 15 | 16
Hypoesthesia (Nervous system disorders) | 24 | 25
Hypertension (Vascular disorders) | 25 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 17
Productive cough (Respiratory, thoracic and mediastinal disorders) | 13 | 7
Constipation (Gastrointestinal disorders) | 50 | 44
Nausea (Gastrointestinal disorders) | 52 | 31
Vomiting (Gastrointestinal disorders) | 24 | 22
Diarrhea (Gastrointestinal disorders) | 30 | 20
Gastroesophageal reflux disease (Gastrointestinal disorders) | 13 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 7
Fever (General disorders) | 33 | 20
Fatigue (General disorders) | 13 | 8
Pain (General disorders) | 14 | 8
White blood cell count decreased (Investigations) | 179 | 161
Neutrophil count decreased (Investigations) | 169 | 158
Platelet count decreased (Investigations) | 98 | 113
AST increased (Investigations) | 14 | 24
ALT increased (Investigations) | 17 | 23
Gamma-glutamyltransferase increased (Investigations) | 4 | 13
Lymphocytes decreased (Investigations) | 15 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT02954172/SAP_000.pdf
  • Study Protocol (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT02954172/Prot_001.pdf